CLINICAL TRIAL: NCT06011174
Title: Validity and Reliability of the Turkish Version of the Post-Stroke Physical Activity Barriers Scale in Patients with Stroke
Status: Completed | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Alper Kemal Gürbüz, research asistant, Kırıkkale University
Other Study IDs: Gurbuz03
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2023-08

CONDITIONS: Stroke; Physical Inactivity
MeSH Terms: conditions — Stroke; Sedentary Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- post-stroke patient: 1. Being 18 years of age or older,
  2. being diagnosed with hemorrhagic or ischemic stroke,
  3. No cooperation and communication problems
  4. Being able to walk independently
  Interventions: Other: survey application

INTERVENTIONS:
Other: survey application — Participants will only be asked to fill out the questionnaires.

SUMMARY:
Stroke is one of the leading causes that negatively affects quality of life. The benefits of regular physical activity are well recognized. Physical activity after stroke may prevent disability and recurrence of stroke. Physical impairments seen after stroke may prevent exercise and limit subsequent recovery. According to a 2016 systematic review updated and published in the Cochrane Library, physical activity programs have positive effects on disability, physical abilities, quality of life, mood and cardiovascular. However, these effects tend to diminish unless the individual's physical activity level is maintained. Therefore, individuals who have had a stroke should be encouraged to exercise. However, it has been reported that most of the patients do not participate in exercise programs as recommended after stroke and there is a decrease in physical activity level. Previous studies have reported that approximately 77% of patients with stroke are sedentary or have low levels of physical activity and also reduced frequency of physical activity. This may be a consequence of the reduced movement speed seen due to severe motor impairments. Interestingly, even those with mild motor impairments, i.e. those walking at speeds above 0.8 m/s and able to participate in community-based exercises, were found to have low levels of physical activity. Therefore, environmental and personal factors can also be barriers to exercise.

Research supports the use of the theoretical model of behavior change developed by Prochaska et al. in physical activity promotion. Individuals are thought to progress through the stages of change at different rates. The concepts of self-efficacy and decision balance (perceived benefits and barriers) are particularly salient for individuals in the pre-thinking and thinking stages. Therefore, identifying and understanding perceived barriers to engaging in physical activity is an important step in creating change in physical activity behaviors. The International Classification of Functioning, Disability and Health defines functioning and disability as multidimensional concepts in which activity, especially physical activity, is influenced by organic and contextual factors. These dimensions often change after stroke and create multiple barriers that may prevent the patient from returning to a physically active lifestyle. Previous studies on barriers to physical activity in stroke survivors have used open-ended questionnaires. When we look at the scales examining exercise and physical activity barriers in the literature, it is seen that they were developed to measure physical activity barriers in the general population and in individuals with chronic conditions. Therefore, the Barriers to Physical Activity After Stroke (BAPAS) scale was developed by Drigny et al. in 2019 to help physicians and therapists identify potential targets for future interventions and optimize clinical follow-up in stroke patients and to assess barriers to physical activity after stroke. The original scale is in French and there is also an English version. Since the scale was recently developed, there is no Turkish version and no version in other languages.

ELIGIBILITY:
Inclusion Criteria:

* 1. Being 18 years of age or older, 2. being diagnosed with hemorrhagic or ischemic stroke, 3. No cooperation and communication problems 4. Being able to walk independently

Exclusion Criteria:

* 1. Having another neurological or orthopedic problem other than stroke that may affect functionality, ambulation and balance 2. Individuals with advanced cardiovascular disease that may prevent physical activity and contraindications for mobilization will not be included in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A standard probability in their use of validity and reliability is unlikely. Generally, it states that at least 3 or 5-10 people should be recruited for each lime substance in lime studies (1,2). For this reason, since the Turkish version of the Post-Stroke Physical Activity Barriers Scale, which consists of 14 items, contains the validity and reliability, it is planned to enroll 70 people with stroke, whose item approach is 5 times higher. Patients coming to Kırıkkale University Faculty of Medicine Physical Therapy and Rehabilitation Hospital will be included in the study.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
the Barriers to Physical Activity After Stroke (BAPAS) SCALE | 10 minute
  The necessary permissions were obtained from the authors of the BAPAS, whose validity and reliability features were to be tested, and the questionnaire was finalized by completing the translation process into Turkish. What is essential in the use of special tools such as scales is to prove the usability of the tool in the sample group to which it will be applied. The first step for this is the translation from the original language to the other language. At this stage, it is ideal to have a good knowledge of the structure of the target language and the original language.
  is to have competent and experienced people do the translation

SECONDARY OUTCOMES:
The Barthel Activities of Daily Living Index (BADLI) | 5 minute
  SURVEY
The Rivermead motor assessment (RMA) | 2 minute
  SURVEY

CONTACTS AND LOCATIONS:
Locations (1):
- Kırıkkale University, Kırıkkale, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes